CLINICAL TRIAL: NCT06027671
Title: Structured Peer-delivered Antiretroviral Therapy (ART) and Reentry Community Strategy to Overcome Barriers to HIV Care Continuity During Community Re-entry From Incarceration in South Africa
Brief Title: Structured Peer-delivered ART and Reentry Community Strategy
Acronym: SPARCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Aurum Institute (Other); Seoul National University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00386911
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Retention in Care
Keywords: Viral Load Suppression; Prison; Transition; Care continuity; HIV

STUDY DESIGN:
Intervention Model Description: This is a hybrid type 1 effectiveness-implementation study to compare care as usual with Full-SPARCS. The investigators will recruit participants from correctional facilities in the Department of Correctional Services (DCS) Gauteng Region, South Africa. Study activities for the intervention arm will be delivered in community venues near to where participants live in Tshwane District, Ekurhuleni District, and City of Johannesburg.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators will perform individual randomization blocked by the correctional facility. Study staff will open numbered envelopes with the allocation following enrolment. Participants will be randomized 1:1 to one of the study arms using sequential envelopes with study arm determination sealed inside. Randomization will be stratified by study site and by sex. The randomization lists for each site/sex combination will be generated through randomly permuted blocks of two, four, and six study assignments with an equal number of group assignments within each block. Study assignments will be masked to staff performing outcome assessments (in-person and telephonic interviews) and the investigators until all outcome data have been collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care-as-usual (CAU) arm (No Intervention): Per DCS routine, at release, participants will receive a referral letter form the DCS health services and, in most cases, will be provided with a 28-day supply of ART.
- Full -SPARCS intervention arm (Experimental): The Full-SPARCS component comprises one individual pre-release session, one individual post-release session, and 12 approximately every-other-week (approximately every two weeks) post-release group sessions extending six months post-release. The SPARCS curriculum is designed to build goal setting, prioritizing, and planning skills during the 12 sessions.
  During each Full-SPARCS session, participants will work with facilitators to set, review, and update personal goals using standardized goal-setting worksheets. These goal sheets will document participant objectives, action steps, timelines, and progress assessments.
  Interventions: Behavioral: Full-SPARCS Intervention

INTERVENTIONS:
Behavioral: Full-SPARCS Intervention — Within 14 days of release, participants will have one-on-one contact with a facilitator to update locator information, continue rapport building, review disclosure plans, provide a reminder of SPARCS logistics, and assign or remind the participant to a SPARCS group based on their location of residence and timing of release (depending on whether this occurred pre-release). Each Full-SPARCS meeting lasts approximately 2 hours, and the sessions occur in a private space in a community venue (e.g., community centre or church).
  Arms: Full -SPARCS intervention arm

SUMMARY:
The overarching goal of this study is to implement a transition community adherence club strategy (Full-SPARCS) for HIV-positive individuals transitioning from correctional to community settings in South Africa. The investigators seek to provide actionable findings to inform policy decisions to contribute to HIV care continuity with this population. The investigators note that effectiveness and scalability often conflict with intervention design; thus, the investigators have proposed testing whether a group approach is effective and the investigators will assess the costs of each component

* To compare the effectiveness of Full-SPARCS to care as usual to achieve HIV RNA suppression 6 months following correctional facility release
* To assess determinants of implementation of Full-SPARCS
* To assess the scalability through costing and cost effectiveness analysis of Full-SPARCS

DETAILED DESCRIPTION:
Background: The South African government has devoted resources towards HIV care in correctional facilities that have resulted in antiretroviral therapy (ART) coverage of >90% and viral load (VL) suppression of >80% among incarcerated people living with HIV (PLWH). However, despite free post-release care, the investigators previously observed that only an estimated 34% were in care three months post-release. The investigators developed, tested, and manualized the Structured Peer-delivered ART and Re-entry Community Strategy (SPARCS) to overcome post-incarceration barriers specific to PLWH returning to the community.8-10 In the investigators randomized controlled pilot of SPARCS, 6-month post-release, continuity of care was 61% in the intervention arm compared to 36% in the usual care arm (p=0.001), demonstrating effectiveness. Full-SPARCS involves 12 biweekly peer facilitator-led group sessions spanning six months post-release. Full-SPARCS is designed to increase self-efficacy, social support, and life skills through facilitated group discussion and curriculum including planning, problem solving, financial literacy, and living with HIV.

Methods: This research study will be conducted in Gauteng Province. Recruitment will occur within correctional facilities of the Department of Correctional Services (DCS) - Modderbee, Kgosi Mampuru II, and Johannesburg. All study interventions will occur following release in either Ekurhuleni District, Tshwane District or Johannesburg District. The study population will be comprised of adult (≥18 years old) corrections inmates, either male or female, with known HIV infection and are receiving ART within the correctional facility and are expected to be released back into the community within 3 months of study enrollment Participants will be randomized 1:1 to either the standard of care or Full-SPARCS using sequential envelopes with study arm determination sealed inside. Study staff will contact participants to ascertain care status and update contact information at one week, one month, three months, six months, nine months, and twelve months from release. Participants assigned to Full-SPARCS will be asked to attend biweekly sessions. Full-SPARCS activities will include - structured curriculum, symptom screening, and routine laboratory monitoring.

Study sample: A total of 400 participants will be randomized to one of the two arms.

Significance: The proposed study is consistent with NIH HIV/AIDS highest priority research and the South African National Strategic Plan on HIV, Tuberculosis (TB), and Sexually Transmitted Infections (STIs) 2017-2022. The research addresses the HIV/AIDS Research Priority of "retention and engagement in these services, and achievement and maintenance of optimal prevention and treatment responses." It also addresses "health disparities" through a focus on recently released inmates, a marginalized population, and fits with the South African National Strategic Plan prioritizing inmates as a key population for HIV services.

ELIGIBILITY:
Inclusion Criteria:

* Incarcerated at one of the participating study enrolment sites, awaiting trial (un-sentenced) and sentenced individuals.
* Diagnosed with HIV and ART at the time of enrolment.
* Anticipated release or trial date within three months of study enrolment.
* Self-report expected to reside in an unrestricted environment within Ekurhuleni, Tshwane, or Johannesburg districts of Gauteng Province and within proximity to one of the SPARCS intervention sites (i.e., within 20km, 45-minute travel time, or two local taxi minibus rides)
* Willing to participate in study post-release follow-up activities and provide contact information for post-release follow-up.

Exclusion Criteria:

* <18 years of age.
* Condition (severe cognitive dysfunction or mental illness) rendering the individual unable to provide informed consent.
* Unable to provide informed consent to participate in the study.
* Assessment by DCS health staff indicating that the individual requires a high intensity of care exceeding that which can be provided in a differentiated model of care setting.
* Not released from the correctional facility during the period of intervention delivery.
* Release to a region outside of Gauteng.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
HIV RNA (viral load) suppression at 6 months | 6 months
  HIV RNA suppression will be defined as a viral load <1000 copies/mL. Participants without viral load data will be assumed to have a viral load >1000 c/mL.

SECONDARY OUTCOMES:
HIV RNA (viral load) suppression at 12 months | 12 months
  HIV RNA suppression will be defined as a viral load <1000 copies/mL. Participants without viral load data will be assumed to have a viral load >1000 c/mL.
Cost-effectiveness | up to 12 months
  Cost effectiveness will be measured by combining standardized data collection tools and an analytic framework developed from prior studies to document and classify resources used (e.g. direct human resources, consumables, capital assets) for all intervention-related activities from design, coordination, to direct delivery.
Percentage of participants receiving ART at 6 months | 6 months
  Participants receiving ART by 6 months post-release.
Percentage of participants receiving ART at 12 months | 12 months
  Participants receiving ART by 12 months post-release.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hoffmann, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- The Aurum Institute - Head office, Johannesburg, Gauteng, South Africa